CLINICAL TRIAL: NCT06646315
Title: Early Versus Standard Care in Cancer Patients in Phase 1 Clinical Trials
Acronym: Psico UFF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Psico UFF1; pr081/20 (Other: Independent review Board - Hospital Universitari de Bellvitge)
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Emotional Adjustment
Keywords: Phase I Clinical Trial; Symptoms control; Psychosocial attention; Emotional distress; Sociofamiliar attention
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early intervention (Experimental): Participants will be assessed using ESAS, ENP and adhoc sociofamiliar questions just before entering their Phase I Clinical Trial (T0). Responses of this assessment will be discussed in a multidisciplinary committee comprised of a palliative physician, a clinical psychologist, a social worker, an oncologist, an hematologist and the Phase 1 Unit referent nurse. According to the patient responses, the committee will decide which needs will be addressed and this will be cited to the corresponding professional (palliative, psychologist and/or social worker) within the following 15 days. The same cycle (assessment - committee - attention) will take place a month after the T0 (T1), and during the following 2 other months (T2 and T3).
  Interventions: Behavioral: Early Intervention
- TAU (No Intervention): Participants will be assessed using ESAS, ENP and adhoc sociofamiliar questions just before entering their Phase I Clinical Trial (T0), one month after (T1), two months after (T2) and three months after (T3).

INTERVENTIONS:
Behavioral: Early Intervention — The Early Intervention consists of the proper attention given to those patients who participate in a Phase I Clinical Trial. The attention will be based on a monthly assessment of their physical, psychological/emotional symptoms and, also their sociofamiliar needs. After having discussed patients's needs in a multidisciplinary committee, each professional (paliiative physician, clinical psychologist and/or wocial orker) will proportionate them the required attention in order to increase their quality of life.
  Arms: Early intervention

SUMMARY:
The goal of this clinical trial is to test de feasibility and effectiveness of and early psychosocial and symptoms attention in cancer patients participating in a Phase I Clinical Trial. The main question it aims to answer is the following: Is an early psychosocial and palliative care attention effective to reduce psychosocial and physical symptoms among participants included in a Phase I Clinical Trial? All participants will answer a questionnaire including the Spanish version of the ESAS (Carvajal, García y Centeno, 2013), the ENP-E (Mateo-Ortega, et al., 2019) and two adhoc sociofamiliar-oriented questions. The assessments will take place just before entering the Phase I Clinical Trial treatment (T0) and one-time per month for three consecutive months (T1-T3). Researchers will compare questionnaire responses of the early-attention group and the control group. The assessment responses from the early-attention group will be monthly discussed in a multidisciplinary committee (just after each assessment) and these will receive the attention according to their needs, either by the palliative professional, the clinical psychologist and/or the social worker. The control group will receive the TAU, by which they will be only followed by their medical professional of reference

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of cancer, under outpatient oncological treatment and follow-up in a Phase 1 clinical trial.
* Having the functional capacity to respond to the study's evaluation measures.

Exclusion Criteria:

* Patients with physical limitations, with severe major depression, significant self-harm ideation, who present symptoms of psychosis or substance abuse, or with difficulty answering the questions of the study's evaluative measures, either due to language issues or due to the presence of cognitive impairment.
* Patients who, at the time of being recruited to start the Phase I clinical trial, are being cared for by one of the following three service: Psycho-oncology, Social Work and Palliative Care, or have been cared for by such services during the last 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Psyhsical symptoms | Three months
  Physical and psychosocial symptoms will be assessed using the ESAS (Edmonton Symptoms Assessment Scale). This scale assesses, using a 10-point Likert scale, the intensity of the following symptoms: pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep, and feeling of wellbeing.
Psychosocial symptoms and needs | Three months
  Psychosocial symptoms will be assessed using the ENP-E (Psychosocial and Spiritual Needs Evaluation Scale). This scale assesses, using a 5-point Likert Scale the following dimensions: mood, sadness, feeling nervous, bearability of the situation, sharing the illness with the family, need for more information about the disease, feeling cared for and supported by family and friends, satisfaction with life, feeling in peace, meaning in life, presence of values and beliefs to cope with the situation, level of well-being. Also, the tool explores economic, family, emotional, spiritual and physical concerns, together to signs of emotional distress.
Sociofamiliar needs | Three months
  Sociofamiliar needs of patients will be assessed using the following ad-hoc questions: In the family unit, are there minors, disabled people or other people who require attention? (e.g.: elderly people with chronic disease).
  Is your habitual residence at such a geographical distance that it entails special needs? Is there a caregiver available? In addition to the disease, do you have any other health problem that limits your day-to-day life? Do you feel capable of sharing the process of the illness with your family? Would you need professional guidance/advice for aspects related to employment procedures, resources, benefits, housing needs, financial aid?

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No